CLINICAL TRIAL: NCT02698020
Title: Oxygen Delivery During General Anesthesia in Newborn Infants: An Open Randomized Controlled Trial of Two Levels of Inspired Oxygen.
Brief Title: Optimized Oxygen Delivery During General Anesthesia in Newborn Infants
Acronym: ANOXneo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANOXneo
Record Dates: First submitted 2016-02-25; First posted 2016-03-03 (Estimated); Last update posted 2018-10-15 (Actual); Status verified 2018-10

CONDITIONS: Oxygen Toxicity; Oxidative Stress
Keywords: Newborn; Anesthesia; Oxygen; Hyperoxia
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): High level of supplemental inspired oxygen
- Room-air (Experimental): Supplemental oxygen only provided if oxygen saturation below target
  Interventions: Procedure: Room-air

INTERVENTIONS:
Procedure: Room-air — Provision of room-air
  Arms: Room-air

SUMMARY:
An open randomized control trial investigating the delivery of two levels of inspired oxygen to newborn infants during general anesthesia.

DETAILED DESCRIPTION:
Eligible infants are infants of less than 44 weeks postconceptional age and without pulmonary disease or demand for supplemental oxygen or assisted ventilation. Control subjects receive current standard of care (anesthesia induction/pre-oxygenation with 80%, maintenance of anesthesia with 40%, and recovery with 80% inspired oxygen). Intervention subjects are maintained on room air throughout the procedure and supplemental oxygen added only if necessary according to the pre-specified oxygen saturation target. Subjects are monitored according to clinical protocols AND with cerebral oximetry (NIRS), transcutaneous measurement of partial pressure of oxygen (pO2), and blood-gas analyses. Blood and urine samples are collected for later analysis of markers for oxidative stress.

ELIGIBILITY:
1. Newborn less than 44 weeks postconceptional age
2. No pulmonary disease, no oxygen requirement, or assisted ventilation
3. No genetic syndrome

Max Age: 4 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-10-10 (Actual)

PRIMARY OUTCOMES:
Transcutaneous and blood-gas pO2 | 30 min
  Area under curve (AUC) and absolute values of pO2

SECONDARY OUTCOMES:
Cerebral Oximetry | 30 min
  AUC of O2 saturation
Atelectasis | 30 min
  Reduced lung compliance as a measure of atelectasis formation
Isoprostane | 4 h
  Level of isoprostanes in blood and urine

CONTACTS AND LOCATIONS:
Overall Officials: Johan Agren, MD, PhD, Principal Investigator — Department of Women's and Children's Health, Uppsala University
Locations (1):
- Uppsala University Hospital, Pediatric anesthesia Unit, Uppsala, Sweden